CLINICAL TRIAL: NCT04993690
Title: A Phase 1 Open-Label Dose Escalation and Expansion Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Preliminary Antitumor Activity of LP-168 in Adult Patients With Relapse or Refractory B-Cell Lymphoma
Brief Title: A Study of LP-168 in Participants With Relapse or Refractory B-Cell Lymphoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Guangzhou Lupeng Pharmaceutical Company LTD. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LP-168-CN101
Record Dates: First submitted 2021-07-27; First posted 2021-08-06 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2024-10

CONDITIONS: B-cell Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell

STUDY DESIGN:
Intervention Model Description: Dose Escalation and determination of MTD; multiple dose levels of LP-168 to be evaluated
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Phase I Dose Escalation (Experimental): Dose Escalation and determination of MTD; multiple dose levels of LP-168 to be evaluated
  Interventions: Drug: LP-168 tablet
- Phase I Dose Expansion A (Experimental): CLL/SLL patients treated with prior regimens.
  Interventions: Drug: LP-168 tablet
- Phase I Dose Expansion B (Experimental): CLL/SLL patients with no prior therapy.
  Interventions: Drug: LP-168 tablet
- Phase I Dose Expansion C (Experimental): MCL patients treated with prior regimens.
  Interventions: Drug: LP-168 tablet
- Phase I Dose Expansion D (Experimental): WM patients treated with prior regimens.
  Interventions: Drug: LP-168 tablet
- Phase I Dose Expansion E (Experimental): MZL patients treated with prior regimens.
  Interventions: Drug: LP-168 tablet

INTERVENTIONS:
Drug: LP-168 tablet — Subjects to take LP-168 orally with 240mL water, without food, Once daily or twice daily

SUMMARY:
This is an open-label, multi-center Phase 1/2 study of oral LP-168 in patients with CLL/SLL and NHL who have failed or are intolerant to standard of care.

DETAILED DESCRIPTION:
This study includes 2 parts: phase 1a (LP-168 monotherapy dose escalation) and phase 1b (LP-168 dose expansion). In phase 1a, patients will be enrolled using an 3+3 design. The starting dose of LP-168 in oral tablet form is 100 mg/day (e.g., 100 mg once daily [QD]). Once the MTD and/or RP2D is identified in phase 1a dose escalation, enrollment will continue to phase 1b dose expansion. Cycle length will be 28 days.

ELIGIBILITY:
Key Inclusion Criteria:

* Per 2017 revised WHO lymphoma classification criteria, subject must have either:

Diagnosed with relapsed or refractory DLBCL or FL and require treatment in the opinion of the Investigator and have received 2 lines SOC.

Diagnosed with relapsed or refractory non-Hodgkin's lymphoma associated with B-cell proliferation (such as CLL\ SLL \ MCL \ MZL \ WM, etc.) in need of treatment in the opinion of the Investigator and have received 1 line SOC.

* Adequate hematologic function.
* Adequate hepatic and renal function.
* Ability to receive study drug therapy orally and willing to receive examinations.
* Willingness of men and women of reproductive potential (defined as following menarche and not postmenopausal [and 2 years of non-therapy-induced amenorrhea] or surgically sterile) to observe conventional and effective birth control.

Key Exclusion Criteria:

* According to the 2017 revised WHO Lymphoma Classification Criteria, patients diagnosed with the following diseases: Burkitt lymphoma or Burkitt-like lymphoma, lymphoblastic lymphoma/leukemia, and post-transplant lymphoproliferative disease(PTLD).
* Prior malignancy (other than the disease under study) within the past 3 years, except for curatively treated basal or squamous cell skin cancer, carcinoma in situ of the cervix or breast cancer.
* Subjects who have received the following treatments within 4 weeks or 5 half-lives before the first dose of LP-168:

Antitumor therapies including myelosuppressive chemotherapy, targeted therapy, biological therapy and/or immunotherapy; Any investigational treatment; Patients who have undergone major surgery, severe trauma or radiotherapy.

* Subjects who have received the following treatments within 2 weeks before the first dose of LP-168:

Steroids or traditional herbal medicine for antitumor purposes; Strong and moderate CYP3A inhibitors and inducers; All drugs that may cause QTc interval prolongation or torsional tachycardia.

* Disease states where clinical manifestations may be difficult to control, including HIV, HBV, HCV, syphilis positive or active bacterial and fungal infections; Disease affects the central nervous system with obvious symptoms; Autoimmune hemolytic anemia or Idiopathic thrombocytopenic purpura. Any gastrointestinal conditions that may severely affect the study drug absorption or pharmacokinetic parameters.
* Subjects who cannot tolerate urine collection, venipuncture, lymph node biopsy, and bone marrow aspiration.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-07-06 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | Up to 24 Months
  Phase 1a
Recommended dose for Phase2 (RP2D) | Up to 24 Months
  Phase Ia/Ib
To evaluate the safety of LP-168 by assessing incidence and severity of treatment-emergent adverse events as determined by CTCAE v5.0 | Up to 24 Months
  Phase Ia/Ib

SECONDARY OUTCOMES:
Overall Response Rate | Up to 24 Months
  To assess the preliminary anti-tumor activity of LP-168 based on overall response rate (ORR) as assessed by investigator and IRC.
Progression Free Survival | Up to 24 Months
  To assess the preliminary anti-tumor activity of LP-168 based on Progression free survival (PFS) as assessed by the Investigator and IRC
Duration of Response | Up to 24 Months
  To assess the preliminary anti-tumor activity of LP-168 based on Duration of response (DOR) as assessed by the Investigator and IRC.
Pharmacokinetics (PK) As Assessed By Maximum Observed Plasma Concentration (Cmax) Of LP-168 | Up to 48 hours post dose
  Phase Ia/Ib
PK As Assessed By Area Under The Plasma Concentration Time Curve From Time 0 To The Time Of The Last Quantifiable Concentration (AUC0-t) Of LP-168 | Up to 48 hours post dose
  Phase Ia/Ib
PK As Assessed By Time To Maximum Observed Plasma Concentration (Tmax) Of LP-168 | Up to 48 hours post dose
  Phase Ia/Ib
PK As Assessed By Terminal Half-life (t1/2) Of LP-168 | Up to 48 hours post dose
  Phase Ia/Ib

CONTACTS AND LOCATIONS:
Overall Officials: Jun Zhu, Study Chair — Peking University Cancer Hospital & Institute
Locations (3):
- China (3):
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong

IPD SHARING:
Plan to Share IPD: No